CLINICAL TRIAL: NCT05305430
Title: A Multi-Center Post-Market Data Collection Protocol to Evaluate the Performance of Synergy Spine Solutions Synergy Disc
Brief Title: Real World Data Collection on the Synergy Cervical Disc
Status: Recruiting | Type: Observational
Sponsor: Synergy Spine Solutions (Industry)
Collaborators: Pacific Clinical Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CP 21-001
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cervical Disc Degeneration
Keywords: degenerative disc; cervical; radiculopathy; myelopathy; motion preservation
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: All patients for whom the decision has been made to have the Synergy Disc implanted at participating investigative centers and give informed consent to participate in the prospective segment of this protocol, per country-specific requirements, will be enrolled in the prospective portion of this protocol.
  Interventions: Device: Synergy Cervical Disc System
- Retrospective: Patients who have previously had a Synergy Spine Solutions Synergy Disc implanted will be eligible for inclusion in the retrospective data collection; a waiver of consent, or informed consent, for retrospective data collection from the medical records of the implanting surgeon will be sought per country-specific regulations as applicable.
  Interventions: Device: Synergy Cervical Disc System

INTERVENTIONS:
Device: Synergy Cervical Disc System — motion preservation disc
  Other Names: Synergy Disc

SUMMARY:
This trial is a real world data (RWD) collection observational study, comprised of both prospective and retrospective arms, that will examine the safety and effectiveness of the Synergy Cervical Disc System in patients with degenerative cervical disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 21 at the time of the surgery.
2. Have had (retrospective cohort) or the decision has been made to have (prospective cohort) the Synergy Disc implanted
3. Skeletally mature patients for reconstruction of the disc from C3-C7 following a single or multiple level discectomy for intractable radiculopathy
4. Intractable radiculopathy and/or myelopathy with at least one of the following producing symptomatic nerve root and/or spinal cord compression: herniated disc and/or osteophyte formation
5. Symptomatic nerve root and/or spinal cord compression documented by patient history (arm or neck pain and/or neurologic deficit) and imaging (CT, MRI, x-rays, etc.)
6. Failed a minimum of 6 weeks conservative treatment
7. Written informed consent given by subject, as applicable.

Exclusion Criteria:

1. Moderate to advanced spondylosis
2. Diagnosis of osteoporosis
3. Active systemic infection or infection at the operative site
4. Pregnancy
5. Marked cervical instability on lateral, coronal, or flexion/extension radiographs
6. Cervical spine condition other than symptomatic cervical disc disease requiring surgical treatment at the involved level
7. Severe pathology of the facet joints of the involved vertebral bodies
8. Previous diagnosis of osteopenia or osteomalacia
9. More than one immobile vertebral level between C1 and T1 from any cause
10. Morbid obesity
11. Currently a prisoner

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both retrospective and prospective study subjects that have cervical degenerative disc disease requiring treatment with the Synergy Spine Solutions Synergy Disc.
  Prospective study cohort: All patients for whom it has been decided that the Synergy Spine Solutions Synergy Disc will be implanted at participating investigative centers and give informed consent to participate in the prospective segment of this protocol.
  Retrospective study cohort: Patients who have previously had a Synergy Spine Solutions Synergy Disc implanted. If required by local regulations, informed consent will be sought and received from the participating patient prior to data collection from the medical records per country-specific regulations.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 12 months
  >15 improvement in NDI score (out of 100) in subjects by 12 mo. post operative compared with baseline
Device Related or Device Procedure Related Adverse Events | 12 months
  Absence of major device related adverse events defined as radiographic failure, neurological failure, or failure by adverse event

SECONDARY OUTCOMES:
Visual Analog (VAS) pain | pre-operative and 6 week, 3 months, 6 months, 12 months, annually post operatively
  Visual analogue scale (VAS) will be used to evaluate pain where a change of at least 20mm will be considered clinically significant. Neck pain as measured on a 100mm VAS at baseline and at each follow-up time-point. Left and Right arm/shoulder pain as measured on a 100mm VAS at baseline and at each follow-up time-point.
Patient Satisfaction | 6 weeks, 3 months, 6 months, 12 months, annually post operatively
  patient completed questionnaire on satisfaction with disc replacement surgery
Nurick's Criteria | pre-operative and 6 weeks, 3 months, 6 months, 12 months, annually post operatively
  disease status characterized by physician at each visit
Odom's Criteria | 6 weeks, 3 months, 6 months, 12 months, annually post operatively
  surgical outcome characterized by physician at each post operative visit
Neurologic Function | 6 weeks, 3 months, 6 months, 12 months, annually post operatively
  maintenance or improvement in neurologic status compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jane M Jacob, PhD, Study Director — Sponsor GmbH
Locations (3):
- Australia (3):
  - Greenslopes Private Hospital, Brisbane, Queensland
  - Dr. Greg Malham, Melbourne, Victoria
  - Spine and Scoliosis Research Associates Australia Ltd, Windsor, Victoria

IPD SHARING:
Plan to Share IPD: No